CLINICAL TRIAL: NCT03257150
Title: Irreversible Electroporation for Locally Advanced Pancreatic Ductal Adenocarcinoma (LEAP TRIAL): A Phase I/II Prospective Trial
Brief Title: A Study of the Use of Irreversible Electroporation in Pancreatic Ductal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEAP
Record Dates: First submitted 2017-08-09; First posted 2017-08-22 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): Single arm trial of irreversible electroporation using the NanoKnife system for locally advanced pancreatic ductal adenocarcinoma.
  Interventions: Procedure: Irreversible Electroporation; Device: NanoKnife System

INTERVENTIONS:
Procedure: Irreversible Electroporation — Irreversible electroporation (IRE) is a process that uses the NanoKnife system to sent electrical currents to a cancer tumor which will disrupt the tumor cell and therefore causing the cell to die. Eligible patients will undergo in situ IRE performed via laparotomy surgery.
Device: NanoKnife System — A system consisting of electrode probes connected to a machine. The probes will be surgically placed around the tumor.

SUMMARY:
This I/II study will evaluate to see how safe and useful irreversible electroporation (also called NanoKnife) is in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
In this phase I/II trial, patients with locally advanced pancreatic ductal carcinoma will be assigned to receive interventional treatment of irreversible electroporation (IRE).

IRE will be performed by laparotomy under general anesthesia in the operating room.

All patients enrolled in the study will have a biopsy at the time of laparotomy. Blood will be collected for regular blood tests and correlative studies at baseline and during the study. Computed tomography (CT) scans will be done at baseline, 4 weeks post treatment, 12 weeks, 24 weeks, and 36 weeks follow up. Quality of Life (QOL) questionnaires will be completed at baseline and during the study. Patients will be given optional consent for storage of any leftover tissue and blood samples for future analysis. Patients will be followed up 4 weeks post treatment, then every 12 weeks until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pancreatic ductal adenocarcinoma (PDAC)
* Age ≥ 18 years
* Locally advanced unresectable primary tumor
* Tumors ≤5 cm in largest dimension at the time of enrollment that is technically amenable to treatment with irreversible electroporation (IRE)
* At least 4 months of combination chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Acceptable organ and bone marrow function
* Life expectancy estimated ≥6 months
* Ability and willingness to sign informed consent form
* Have a measurable primary tumor at the time of study enrollment
* Suitable and fit to undergo general anesthetic and laparotomy
* Women of child-producing potential must agree to use effective contraceptive methods prior to study entry, during study participation, and for at least 30 days after the last administration of study medication.

Exclusion Criteria:

* Stage IV (i.e. metastatic) PDAC
* Have a cystic subtype PDAC of the pancreas
* Previous local treatments for locally advanced PDAC including IRE or radiotherapy
* Recent or concurrent cancer, that is distinct from PDAC in primary site/histology, except cervical carcinoma in situ, localized prostate cancer, treated basal cell carcinoma, superficial bladder tumours (Ta, Tis & T1) and those that can be permitted with sufficient clinical justification confirming patient safety to undergo the procedure per Principle Investigator and is in the best interest of the patient. Cancer curatively treated ≥3 years prior to entry is permitted.
* Prior chemotherapy within 3 years of diagnosis of PDAC. Chemotherapy for PDAC is permitted
* Direct invasion of locally advanced PDAC into the stomach or duodenum
* Metallic biliary stent that cannot be substituted with a plastic stent
* Allergy to computed tomography (CT) or magnetic resonance imaging (MRI) contrast that cannot be safely managed with premedication which preclude assessment and/or surveillance of PDAC
* History of cardiac disease (including, but not limited to: congestive heart failure, active coronary artery disease, uncontrolled hypertension)
* Any active major medical illnesses of the respiratory or immune system, or other conditions that may affect patient's ability to tolerate general anesthesia and IRE therapy on this trial
* History of solid organ transplantation or collagen vascular disease
* Medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Pregnant or breast feeding women
* Pre-menopausal women unwilling to take a pregnancy test
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g.: infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.)
* History of human immunodeficiency virus (HIV) infection
* Progression of the primary lesion as judged by the Investigator
* Working knowledge of English is a must in order to complete the quality of life questionnaires being administered in this study. Patients who do not meet this requirement will be exempt from the quality of life assessments but remain eligible for all other components of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Adverse event rate | 30 days post IRE or index hospitalization
Overall survival rate | Date of IRE treatment to the date of death, up to 2 years

SECONDARY OUTCOMES:
Progression-free survival rate | IRE treatment to the date of documented disease progression or death, up to 2 years
Overall survival rate of disease | Date of disease diagnosis to date of death, up to 2 years
Progression-free survival rate of disease | Date of disease diagnosis to date of death, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gallinger, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No